CLINICAL TRIAL: NCT04360525
Title: Different Clinicopathological Features of Non-Elderly Sigmoid Volvulus Patients
Status: Completed | Type: Observational
Sponsor: Dr. Ersin Arslan Education and Training Hospital (Other Government)
Collaborators: Inonu University (Other)
Responsible Party: Principal Investigator, Ufuk Uylas, Specialist, Dr. Ersin Arslan Education and Training Hospital
Other Study IDs: 18042020
Record Dates: First submitted 2020-04-18; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Pathology
Keywords: dolichocolon; volvulus; sigmoid; Parkinson; mental retardation; Hirschsprung's disease
MeSH Terms: conditions — Intestinal Volvulus; Intellectual Disability; Hirschsprung Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Elderly patients: Elderly patients (60≤ age) with sigmoid volvulus
  Interventions: Other: Reasons
- Young patients: Young patients (<60 age) with sigmoid volvulus
  Interventions: Other: Reasons

INTERVENTIONS:
Other: Reasons — Causes of sigmoid volvulus

SUMMARY:
Sigmoid volvulus is frequently seen in male patients over 60 years old. In the sigmoid volvulus <60 age groups, the male/female ratio is close to each other. If sigmoid volvulus develops in <60 age groups, it is more likely to be another underlying organic pathology.

DETAILED DESCRIPTION:
Sigmoid volvulus is frequently seen in male patients over 60 years old. Here, the investigators aimed to investigate the causes of sigmoid volvulus developing in patients under 60 years of age. Patients diagnosed with sigmoid volvulus between 2009 and 2018 were retrospectively screened. The patients were divided into two as under 60 years old and above. The co-morbidity, mortality, morbidity, complications, age and gender data of the patients were analyzed. In the sigmoid volvulus <60 age groups, the male/female ratio is close to each other. If sigmoid volvulus develops in <60 age groups, it is more likely to be another underlying organic pathology.

ELIGIBILITY:
Inclusion Criteria:

* Sigmoid volvulus patients under the age of 60
* Sigmoid volvulus patients at the age of ≥60

Exclusion Criteria:

* Lack of data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who were treated for the sigmoid volvulus between 2009 and 2018 at Inonu University General Surgery Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-18 (Actual)

PRIMARY OUTCOMES:
Mortality | up to three months
  Elderly and young patients mortality
Morbidity | up to three months
  Elderly and young patients morbidity

CONTACTS AND LOCATIONS:
Overall Officials: ufuk uylas, Specialist, Principal Investigator — Dr. Ersin Arslan Training and Resource Hospital
Locations (1):
- Dr. Ersin Arslan Training and Resource Hospital, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided